CLINICAL TRIAL: NCT05928104
Title: Optimising Pharmacist-led Medication Reviews in Primary Care (OPen): a Qualitative Study to Co-design and Test an Optimised Medication Review for Patients With Long-term Conditions.
Brief Title: Optimising Pharmacist-led Medication Reviews in Primary Care
Acronym: OPen
Status: Completed | Type: Observational
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 313644
Record Dates: First submitted 2023-06-12; First posted 2023-07-03 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-06

CONDITIONS: ALL, Adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Medication Review

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Medication review — Pharmacist-led medication review in primary care using a co-designed document

SUMMARY:
An increasing number of people are diagnosed with long-term conditions and are prescribed medicines to manage these conditions. Medication reviews (MRs) are used to optimise medicines, improve health outcomes, and decrease medicines related problems.

Although medication reviews are widely used in health care settings, there has not been a dramatic change in the the rate at which patients experience poor medicines outcomes such as adverse drug reactions and hospitalisations.

This research wants to understand how medication reviews by pharmacists are delivered in GP surgeries and community pharmacies. The research team plans to test a co-designed document, which outlines what pharmacists should do in a MR, in a small number of GP surgeries, on a limited number of patients.

Pharmacists and patients who have used this document will be interviewed to understand their thoughts and feelings about the process.

DETAILED DESCRIPTION:
Approximately 15 million people in England have a long-term condition (LTC) or chronic disease, such as heart disease, asthma, diabetes, for which there is currently no cure. Long-term conditions are mostly managed by medicines with 1.12 billion prescription items dispensed in England in 2019 at a total cost of £9.08 billion. Recent government reports have identified that prescribing too many or inappropriate medicines can lead to more medicines related problems and poor patient outcomes, such as drug interactions, adverse drug reactions, reduced quality of life, and hospitalisations.

Medication reviews are used to support patients with their medicines and to reduce the risk of over and inappropriate prescribing. Desired outcomes for medication reviews include optimising medicines, improving health outcomes, and decreasing medicines related problems. It has become more common for medication reviews to be used by doctors, nurses, and pharmacists in the last ten years, but the rate at which patients experience poor medicines outcomes such as adverse drug reactions and hospitalisations because of medicines use has not changed much in this time.

Pharmacists are considered to be medicines experts, so many organisations are encouraging them to be involved with the delivery of medication reviews. Pharmacists currently undertake various types of medication reviews in general practitioner (GP) surgeries, Primary Care Networks (PCN), and community pharmacies.

When interventions are introduced to address problems such as overprescribing, it is important to better understand how they have been designed and delivered. The Medical Research Council (MRC) has provided guidance on the process evaluation of complex interventions (of which medication reviews are an example).

This states that the key steps in evaluating complex interventions are:

* Understanding how and what is delivered Understanding how the intervention produces change
* Understanding how context affects implementation and outcomes

To understand the evidence for pharmacist-led medication reviews, a scoping review was undertaken with the aim of describing the existing, extensive literature in this field. This scoping review identified numerous systematic reviews that included a significant quantity of primary research from a wide range of countries. It concluded that overall evidence for effectiveness for medication reviews is uncertain (no strong evidence for or against their effect on patient outcomes). In addition, it identified that most reviews did not describe in depth what is delivered and how the intervention produces change. Therefore, it is difficult to know, from the existing systematic review literature, which elements of the medication review are likely to benefit the patient and the health service.

As a follow-up to this scoping review a systematic review was undertaken to explore what is delivered (the core components of pharmacist-led medication reviews), and whether and how they link to outcomes in different contexts. In addition to extracting data about context, implementation, outcomes, and mechanisms of impact (how intervention produces change), this systematic review also extracted information about actions that affect patients' medicines taking behaviour and implementation strategies (activities that describe how an intervention was delivered).

The output from the systematic review was a draft programme theory. A programme theory describes how an intervention is expected to lead to its effects and under what conditions. The programme theory for pharmacist-led medication reviews shows how the intervention may achieve patient and health service outcomes

The literature reviews have established what has been reported in previous studies, and the evidence for pharmacist-led medication reviews. The next step is to find out what is happening in practice. The current GP and community pharmacy contracts provide some guidance to the provision of medication reviews. However, these documents lack details on why elements have been included and how they will benefit the patient. Focus groups with patients and practitioner (pharmacists, GPs and practice nurses) were undertaken to establish what is happening is practice and the key uncertainties (unknown or incomplete essential details relating to the content and implementation of medication reviews) are. The results from the focus groups, combined with the outcomes from the systematic review were used to design an optimised, evidence-informed pharmacist-led medication review, with the help of stakeholders, such as pharmacists, patients, and GPs.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years

Due for a medication review by the practice pharmacist

Effectively communicate in English

Provide informed consent

Exclusion Criteria:

* Have no access to telephone/ internet

Recently received a medication review

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the general practice sites that are recruited to participate in the study. These sites will be located in Norfolk, Suffolk and North East Essex
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Patient feasibility and acceptability | 3 months
  Patients will be interviewed to assess their thoughts and feelings after receiving the medication review
Pharmacist feasibility and acceptability | 3 months
  Pharmacists will be interviewed to assess their thoughts and feelings after delivering medication reviews using the service specification

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Toftwood surgery, Dereham, Norflok
  - North Elmham surgery, Dereham, Norfolk
  - Sheringham Medical Practice, Sheringham, Norfolk

IPD SHARING:
Plan to Share IPD: No